CLINICAL TRIAL: NCT00047749
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Intrathecal Ziconotide in Adults With Severe Chronic Pain
Brief Title: Prialt (Ziconotide) In Severe Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elan Pharmaceuticals (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ELN92045-301
Record Dates: First submitted 2002-10-16; First posted 2002-10-17 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Pain
Keywords: pain; ziconotide; Prialt; intrathecal; Synchromed
MeSH Terms: conditions — Pain | interventions — ziconotide

INTERVENTIONS:
Drug: Prialt (ziconotide)

SUMMARY:
The purpose of this study is to understand the effects of intrathecal ziconotide (an experimental pain medication) when the dose is slowly increased over a 3-week period in patients with severe chronic pain. During the weaning phase, the study will also gather information about switching from other intrathecal or IT medication (slowly pumped directly into the space around the spine) to other systemic pain medication (by mouth or through the skin using a patch). After being weaned off current IT medication, patients will be placed on IT ziconotide or placebo (non-active substance) as well as being allowed a stable dose of systemic pain medications.

Patients who complete this study may be eligible for long-term ziconotide therapy via extension protocol ELN92045-352.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read, understand, and voluntarily sign the Institutional Review Board (IRB) approved, written informed consent document prior to the performance of any study-specific procedures;
* Patient must be male or female at least 18 years of age;
* Patient must have severe chronic pain for whom IT therapy is warranted;
* Patient must be willing and able to comply with the protocol, and able to maintain the Patient Daily Diary for Opioid Consumption;
* Patient must have an implanted programmable SynchroMed® Infusion System in place for the treatment of chronic pain;
* Female patients of childbearing age agree to use adequate, appropriate contraceptive methods.

Males and their partner(s) of childbearing age must use adequate, appropriate contraceptive methods.

Exclusion Criteria:

* Patient is pregnant or lactating;
* Patient has been on an investigational drug other than ziconotide or device within 30 days prior to the initiation of the study drug;
* Patients with a known hypersensitivity (allergy) to ziconotide or any of the excipients (other compounds) in the formulation;
* Patient has a condition that would contraindicate the use of IT analgesia, including the presence of infection at the microinfusion injection site (where the needle is inserted in your abdomen to fill the pump with medication), uncontrolled bleeding diathesis (tendency for bleeding) and spinal canal obstruction that impairs circulation of Cerebral Spinal Fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2002-08; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Tennesee Valley Pain Consultants - Center For Pain Management, Huntsville, Alabama
  - The Pain Center, Northport, Alabama
  - Outcomes Research International, Tucson, Arizona
  - The RC Goodman Pain Institute: Clinical Research, Fort Smith, Arkansas
  - Hot Springs Mercy Pain Clinic, Hot Springs, Arkansas
  - Innovative Spine Care, Little Rock, Arkansas
  - Advanced Pain Medicine, Bakersfield, California
  - Advanced Pain Institute, Duarte, California
  - UCSD Medical Center, Thornton Hospital, La Jolla, California
  - Abaci and Massey Pain Center, Los Gatos, California
  - UCSF Pain Management Center, San Francisco, California
  - Pain Care Specialists, Colorado Springs, Colorado
  - Clinical Pharmacology Services, Inc., Tampa, Florida
  - Georgia Medical Research Institute, Marietta, Georgia
  - Rush Presbyterian - St. Luke's Medical Center, Chicago, Illinois
  - University of Kentucky, Dept Anesthesiology, Lexington, Kentucky
  - Johns Hopkins Hospital, Division of Pain Management, Baltimore, Maryland
  - Arnold Pain Management, Boston, Massachusetts
  - Edina Medical Pain Center, Edina, Minnesota
  - Research Medical Center - Pain Institute, Kansas City, Missouri
  - Yellowstone Medical Center East, Billings, Montana
  - Huntington Center for Pain Treatment, Huntington, New York
  - Weill Medical College of Cornell University, New York, New York
  - Medical Pain Management of Central NY, Syracuse, New York
  - Center For Clinical Research, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Pain Institute of Tulsa, Tulsa, Oklahoma
  - Pain Consultants of Oregon, Eugene, Oregon
  - Legacy Holladay Park Medical Center, Portland, Oregon
  - Penn State University Hospital, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Advanced Clinical Concepts, Temple, Pennsylvania
  - Neurosurgery Foundation, Providence, Rhode Island
  - MUSC, Neurological Surgery, Charleston, South Carolina
  - Methodist Comprehensive Pain Institute, Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Texas Tech University HSC, Lubbock, Texas
  - Consultants in Pain Research, San Antonio, Texas
  - Alpine Pain and Addiction Medicine, Salt Lake City, Utah
  - Advanced Pain Management and Rehabilitation, Virginia Beach, Virginia
  - University of Washington Medical Center - Pain Center, Seattle, Washington
  - Center for Pain Relief, Charleston, West Virginia
  - Cardinal Clinical Research Center, Cudahy, Wisconsin

REFERENCES:
- See also: Ziconotide in severe chronic pain (search using ziconotide) — http://www.centerwatch.com